CLINICAL TRIAL: NCT00213057
Title: A Randomized, Placebo-controlled, Double-blind Trial to Assess Expanded Safety and Acceptability of Carraguard™ (PC-515) Vaginal Gel Among Heterosexual Couples in Chiang Rai
Brief Title: Safety and Acceptability of Carraguard™ Among HIV-negative Couples in Thailand
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Ministry of Health, Thailand (Other Government); Chiang Rai Public Health Office (Other Government); Chiang Rai District Health Office (Other Government); Chiang Rai Municipal Health Office (Other Government); Chiang Rai Hospital (Other); Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Population Council #270; CDC Protocol #2968
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections; Chlamydia Trachomatis; Nesseria Gonorrhea; Trichomonas Vaginitis; Syphilis
Keywords: Microbicides; HIV prevention; sexually transmitted infections; carrageenan; sero-concordant couples; HIV Seronegativity; HIV
MeSH Terms: conditions — HIV Infections; Trichomonas Vaginitis; Syphilis; Sexually Transmitted Diseases

INTERVENTIONS:
Drug: Carraguard (PC-515)

SUMMARY:
The primary aims of the study were to assess the safety and acceptability of Carraguard applied vaginally prior to sexual intercourse for six months in both women and men; and to examine several dimensions of acceptability. Secondary aims were to gauge reactions to a non-contraceptive microbicide, to assess use dynamics among Thai couples and to observe preliminary indications of sexually transmitted infections and reproductive tract infections averted.

The hypothesis was that Carraguard would cause little or no significant irritation, including lesions; and that women and men would find Carraguard acceptable.

DETAILED DESCRIPTION:
Carraguard™ (PC-515), the Population Council's lead candidate microbicide, was tested in a triple-masked, randomized, placebo-controlled trial fielded in one site in Chiang Rai, northern Thailand. The primary aims of the study were to assess Carraguard's safety (toxicity) in both men and women - including signs of local irritation, such as itching or burning; changes in vaginal flora (women); and incidence of abnormal external genital, vaginal (women), and cervical findings (women) - when applied vaginally prior to intercourse for 6 months; to evaluate acceptability; to gauge men's and women's reactions to a non-contraceptive microbicide; and to explore microbicide use dynamics in a Thai population.

Secondary aims were to investigate sexually transmitted infections averted - including HIV, C. trachomatis, N. gonorrhoeae, T. vaginalis, and T. pallidum (preliminary indications) in men and women; bacterial vaginosis and candidaisis in women; and balanitis in men; and effect on cervical cytology.

ELIGIBILITY:
Inclusion Criteria:

* · In good health,

  * Aged 18 years or older,
  * Resident for at least 1 year; planning to stay for at least 12 months,
  * HIV-seronegative and free of all other STD at initial screening exam,
  * No reported sex partners other than current partner for prior year and and not planning on having any other sex partners for the duration of the study,
  * Not using condoms routinely (>25% of the time) in the prior year
  * Willing and able to comply with the study protocol (including being tested for HIV, learning the results, agreeing to partner notification if a curable STD is diagnosed, and undergoing clinical evaluations),
  * Able to achieve a score of 80% or better on true-false test of key study concepts, and
  * Able to give informed consent.
  * Planning to have vaginal sexual intercourse together on average at least once per week during the next six months.

Exclusion Criteria:

* · Pregnant or desire to become pregnant at time of study participation,

  * Delivered or aborted a pregnancy within the six weeks prior to screening,
  * Male sex partner known at enrollment to be HIV positive,
  * History of surgery on external genitalia, vagina or cervix in the six weeks prior to screening,
  * Recent history of non-menstrual vaginal bleeding with intercourse,
  * Clinically detectable genital abnormality (including presence of warts, or a structural or congenital abnormality),
  * Genital epithelial disruption; men/women with healed lesions (intact epithelium) will be eligible,
  * Untreated symptomatic bacterial vaginosis or candidiasis. Women with asymptomatic BV or yeast may be enrolled. Women with treated symptomatic BV or candidaisis may be enrolled once no longer symptomatic. Women with signs or laboratory evidence of BV or candidaisis may be enrolled if they are asymptomatic. Women with symptoms of vaginal infection may be enrolled only if their enrollment visit stat laboratory evaluation is negative for BV, candidaisis or trichomoniasis,
  * Presence of balanitis. Men with resolved balanitis (e.g. through treatment) will be eligible,
  * Abnormal Pap smear (Class II or above),
  * History of sensitivity/allergy to latex,
  * Concurrent participation in another trial of a vaginal product,
  * Injection of recreational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2001-06 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Safety (toxicity/local irritation): Genital exam and interview for signs and symptoms, 14-days after enrollment and monthly thereafter for 6 months; testing for bacterial vaginosis and candida (women) and balanitis (men) monthly.
Acceptability: Interview about gel use to assess compliance (monthly) and acceptability (quarterly).

SECONDARY OUTCOMES:
Preliminary effectiveness: Swabs taken from women an urine specimens collected from men to test for sexually transmitted infections - gonorrhea, chlamydia, trichomoniasis (monthly) and for genital ulcer disease, if ulceration was detected; blood drawn

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Blanchard, MSc, Principal Investigator — Population Council
Locations (1):
- Chiang Rai Health Club, Chiang Rai, Thailand